CLINICAL TRIAL: NCT04563949
Title: Clinical Practice Utility Study to Assess DermTech's Non-Invasive Pigmented Lesion Assay to Detect and Track Lesions for Suspected Melanoma and to Determine Outcomes for up to 2 Years
Brief Title: DermTech's Non-Invasive Pigmented Lesion Assay to Detect and Track Lesions for Suspected Melanoma and to Determine Outcomes for up to 2 Years
Acronym: TRUST
Status: Completed | Type: Observational
Sponsor: DermTech (Other)
Responsible Party: Sponsor
Other Study IDs: 17-02
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2020-09

CONDITIONS: Melanoma Detection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA extracted from DermTech's PLA assay for gene expression observed in melanoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PLA-: PLA- initially and repeat testing 1-2 years later
  Interventions: Other: Repeat Testing
- PLA+: Not eligible for the study

INTERVENTIONS:
Other: Repeat Testing — Repeat Testing with the PLA will be conducted
  Groups: PLA-

SUMMARY:
This is a multi-center, sample collection study to follow clinically suspicious lesions to determine the outcome including surgical biopsy, removal, monitoring, etc. for up to 2 years after lesion identification. Subjects who had, or will have a DermTech Pigmented Lesion Assay completed on a lesion suspected of being melanoma are eligible for the study. Based on historical data, an expected melanoma rate of approximately 5% to 10% is anticipated.

DETAILED DESCRIPTION:
This is a multi-center, sample collection study to follow clinically suspicious lesions to determine the outcome including surgical biopsy, removal, monitoring, etc. for up to 2 years after lesion identification.

Subjects will be consented and enter the trial to have their suspicious lesion(s), biopsied via DermTech's adhesive patch biopsy and assessed with DermTech's non-invasive PLA, and followed up to 2 years per standard of care. Lesions must be photographed and/or the site of the lesion anatomically defined to permit follow-up of the lesion(s) and lesional site(s) during future visits.

Subjects will be followed per standard of care for lesion biopsy, excision, treatment and/or monitoring. Other than DermTech's non-invasive PLA of the lesion(s) no other study procedures will be performed and subjects will be treated according to the standard of care. The subject's medical management team should use standard of care, visual assessment changes (i.e., "ABCDE") and physician judgment for suspicious lesion characterization and monitoring when planning the subject's course of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females the treating physician chose to use the PLA on;
2. Presence of a lesion(s) that is suspicious for melanoma and a candidate for surgical biopsy that was previously biopsied with DermTech's adhesive patch biopsy and assessed via PLA;
3. Willing to permit subsequent PLA assays to be performed on suspicious lesions;
4. Willing to follow standard of care treatment for the lesion(s) as determined by the treating physician;
5. Subjects must be able to complete study visits required by the protocol (subject is not planning to relocate or travel thus prevent attendance at future study visits; and
6. Willing to provide informed consent to participate in this trial.

Exclusion Criteria:

1. Has confirmed melanoma or a suspicious lesion that required a surgical biopsy or excision prior to the intial PLA on that lesion of interest;
2. Has an ulcerated or bleeding lesion that could cofound the PLA results;
3. Has a suspicious lesion(s) in an area that was previously surgically biopsied;
4. The lesion(s) is on the palms, mucosal surface, or other area where adhesive patch biopsies cannot be performed;
5. Has an allergy to tape or latex rubber;
6. Receipt of any investigational drug therapy within four weeks of study enrollment, or concurrent participation in another interventional clinical study deemed by the treating physician to potentially influence this study; and
7. Documented substance abuse, any other significant medical condition or laboratory result that would indicate an unreasonable risk to the subject or potential interference with study procedures, or would negatively affect the patient's reliability and compliance with the study schedule of events. -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who had a DermTech PLA completed on a lesion suspected of being melanoma are eligible for the study. Based on historical data, an expected melanoma positivity rate of 5%-10% is anticipated.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects without surgical biopsy | approximately up to 24 months
  The proportion of subjects who exit the study without surgical biopsy out to approximately up to 24 months ± SOC

SECONDARY OUTCOMES:
Results of PLA results compared to biopsy | approximately up to 24 months
  Expression of genes during the 2-year study. The association of gene expression and algorithm values with melanoma versus non-melanoma will be examined using clinical performance indicators negative predictive value with their respective 95th percentile confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
All samples received have been de-identified with a study and subject specific number.

REFERENCES:
- [Background] Ferris LK, Jansen B, Ho J, Busam KJ, Gross K, Hansen DD, Alsobrook JP 2nd, Yao Z, Peck GL, Gerami P. Utility of a Noninvasive 2-Gene Molecular Assay for Cutaneous Melanoma and Effect on the Decision to Biopsy. JAMA Dermatol. 2017 Jul 1;153(7):675-680. doi: 10.1001/jamadermatol.2017.0473. PMID 28445578
- [Background] Gerami P, Yao Z, Polsky D, Jansen B, Busam K, Ho J, Martini M, Ferris LK. Development and validation of a noninvasive 2-gene molecular assay for cutaneous melanoma. J Am Acad Dermatol. 2017 Jan;76(1):114-120.e2. doi: 10.1016/j.jaad.2016.07.038. Epub 2016 Oct 1. PMID 27707590